CLINICAL TRIAL: NCT02617693
Title: Jom Mama Project - Pre-pregnancy Intervention to Reduce the Risk of Diabetes and Prediabetes
Brief Title: Development of Pre-pregnancy Intervention to Reduce the Risk of Diabetes and Prediabetes
Acronym: Jom Mama
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INS-4186; U1111-1160-2987 (Other: WHO)
Record Dates: First submitted 2015-11-18; First posted 2015-12-01 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Other)
  Interventions: Other: standard antenatal care
- Life style intervention (Experimental)
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Behavioral: lifestyle intervention — Evaluation of lifestyle intervention combining behavioural change councelling and utilisation of E-health platform. The intervention consists of a combination of behaviour change counselling and support through six contact-points with CHPs (community health promoter) and access to a personalised mobile application.
  Arms: Life style intervention
Other: standard antenatal care — Standard of care for pre-pregnancy health. Subjects will be reminded of their endpoint measurement visit towards the end of the intervention period through a phone call.
  Arms: Standard of care

SUMMARY:
This study is conducted in Asia. The aim of this study is to assess the efficacy of a pre-pregnancy life style intervention to reduce the risk of diabetes and prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Nulliparity
* Not pregnant at the time of signing informed consent
* Own a smartphone with either Android system version 4.1 and above or iOS system 7.0 and above with internet access

Exclusion Criteria:

* Female subject undergoing treatment for type 1 or 2 diabetes mellitus
* Subjects not residing in the district of Seremban

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2017-12-09 (Actual); Study Completion 2017-12-09 (Actual)

PRIMARY OUTCOMES:
Difference in waist circumference | Months 0-8

SECONDARY OUTCOMES:
Change in BMI (Body Mass Index) | Month 0, Month 8
Change in waist-to-height ratio (WHtR) | Month 0, Month 8
Change in waist-to-hip ratio | Month 0, Month 8
Change in weight | Month 0, Month 8
Change in HbA1c (Glycosylated haemoglobin)) | Month 0, Month 8
Change in the fasting lipid profile (total cholesterol [TC], low density lipoprotein cholesterol[LDL-C], high density lipoprotein cholesterol[HDL-C], triglycerides [TG]) | Month 0, Month 8
Change in blood pressure (SBP (systolic blood pressure) and DBP(diastolic blood pressure)) | Month 0, Month 8
Change in the level of health literacy, as measured by the European Health Literacy Survey Questionnaire (HLC-EU-Q) | Month 0, Month 8
Change in dietary intake, as measured by the Frequency Food Questionnaire (FFQ) that is used in National Health Surveys in Malaysia | Month 0, Month 8
Change in dietary intake, as measured by a Frequency Food Questionnaire (FFQ) | Month 0, Month 8
Change in physical activity and sedentary behaviour, as measured by the International Physical Activity Questionnaire (IPAQ) used in National Health Surveys in Malaysia | Month 0, Month 8
Change in stress levels, as measured by the Depression Anxiety and Stress Scale 21-items (DASS-21) used in National Health Surveys in Malaysia | Month 0, Month 8

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seremban, Negeri Sembilan, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk.com

REFERENCES:
- [Derived] Skau JK, Nordin AB, Cheah JC, Ali R, Zainal R, Aris T, Ali ZM, Matzen P, Biesma R, Aagaard-Hansen J, Hanson MA, Norris SA. A complex behavioural change intervention to reduce the risk of diabetes and prediabetes in the pre-conception period in Malaysia: study protocol for a randomised controlled trial. Trials. 2016 Apr 27;17(1):215. doi: 10.1186/s13063-016-1345-x. PMID 27117703
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com